CLINICAL TRIAL: NCT00161863
Title: Open-label Safety Study of FSME-IMMUN NEW in Healthy Children and Adolescents Aged 1 to 15 Years
Brief Title: Safety Study of FSME-IMMUN NEW in Healthy Children and Adolescents Aged 1 to 15 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 209
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Tick-borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: FSME-IMMUN NEW 0.25 ml

SUMMARY:
The purpose of this study is to investigate the safety of five consecutive lots of FSME-IMMUN NEW in healthy volunteers. The main criterion for investigation is the fever rate after the first vaccination in three different age classes. The immunogenicity of 0.25 ml FSME-IMMUN NEW has been demonstrated in previous clinical studies in children; therefore, in the present study, immunogenicity was investigated in a subgroup only.

ELIGIBILITY:
Inclusion Criteria:

Male and female children and adolescents will be eligible for participation in this study if:

* they are aged 1 year (from the 1st birthday) to < 16 years (to the last day before the 16th birthday);
* they are clinically healthy, (i. e. the physician would have no reservations vaccinating with FSME-IMMUN NEW outside the scope of a clinical trial);
* their parents/legal guardians understand the nature of the study and agree to its provisions;
* written informed consent is available from both parents/legal guardians,
* for Germany/Austria: additional written informed consent is available for children older than 8 years
* they or their parents/legal guardians agree to keep a volunteer diary.

For safety reasons, female volunteers who have reached sexual maturity at study start have to meet the following additional inclusion criteria:

- negative pregnancy test at study entry;

Exclusion Criteria:

Children and adolescents will be excluded from participation in this study if they:

* have a history of any TBE vaccination;
* have a history of TBE infection;
* have a history of allergic reactions to one of the components of the vaccine;
* suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids, chemotherapeutics) that can be expected to influence immunological functions;
* are known to be HIV positive (a special HIV test is not required for the purpose of the study);
* have received banked blood or immunoglobulins within one month of study entry;
* have a history of vaccination against yellow fever and/or Japanese B-encephalitis;
* suffer from hemorrhagic diathesis;
* are participating simultaneously in another clinical trial;
* if female: are pregnant or breastfeeding.

Volunteers who meet the inclusion/exclusion criteria, but have a febrile illness (body temperature > 38°C) at the scheduled time of vaccination, will not be vaccinated before their body temperature returns to normal.

Volunteers who have received any other vaccination within 4 weeks prior to visit 1 will not be vaccinated until an interval of 4 weeks has passed. In this case visit 1 will take place separately.

If volunteers have received antipyretics within 4 hours prior to the intended TBE vaccination, the vaccination should be performed at a later time.

Volunteers who have a positive TBE antibody value prior to the first vaccination will be excluded from the statistical analysis of the primary endpoint.

Ages: 1 Year to 15 Years | Sex: All
Age Groups: Child
Dates: Start 2002-09; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter BioScience
Locations (8):
- Grieskirchner Strasse 17, Wels, Austria
- Germany (3):
  - Marktplatz 3, Bad Saulgau
  - Solothurner Strasse 2, Heilbronn
  - Hauptstraße 240, Kehl
- Poland (4):
  - Wojewodzki Szpital Dziececy oddz. Obserwacyjno-Zakazny, Kielce
  - Szpital Jana Pawla II Odz. Neuroinfekcji, Krakow
  - Samodzielny Publiczny ZOZ Oddzial Dzieciecy, Lubartów
  - PANTAMED sp.z.o.o., Olsztyn